CLINICAL TRIAL: NCT00431769
Title: A Phase II, Open-Label Trial Using Velcade for ReTreatment of Multiple Myeloma Subjects Following an Initial Response to Velcade
Brief Title: An Efficacy and Safety Study of Bortezomib Re-treatment in Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR010519; 26866138MMY2036 (Other: Janssen-Cilag International NV); 2005-005819-26 (EudraCT Number)
Record Dates: First submitted 2007-02-02; First posted 2007-02-06 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Bortezomib; Dexamethasone; VELCADE
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bortezomib (Experimental)
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib — Bortezomib will be given intravenously (into a vein) twice weekly, on Days 1, 4, 8 and 11 and then a 10-day (Days 12 to 21) rest period, of each 3-week cycle for up to a total of 8 cycles. The initial bortezomib dose is 1.0 or 1.3 milligram per meter square (mg/m^2) depending on the previous bortezomib-based treatment, up to a maximum dose of 1.3 mg/m^2. Participants will receive bortezomib in combination with or without dexamethasone, in accordance with the standard of care. The median total dose of dexamethasone per cycle ranges from 120 mg (Cycle 7) to 160 mg (Cycles 1 to 6 and 8).

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of bortezomib in participants with multiple myeloma who have previously responded to a bortezomib based therapy.

DETAILED DESCRIPTION:
This is an Open-Label (all people know the identity of the intervention), non-randomized, multicenter (when more than one hospital or medical school team work on a medical research study), single arm study to evaluate the safety and efficacy of bortezomib in participants with multiple myeloma (cancer of the types of cells normally found in bone marrow) who have previously responded to a bortezomib based therapy. Participants will be non-randomly assigned to single group bortezomib. Participants will be treated with bortezomib alone or in combination with another drug (dexamethasone). Bortezomib will be given intravenously (i.v. [into a vein]) twice Weekly, on Days 1, 4, 8 and 11 of each cycle followed by a 10-day (Days 12 to 21) rest period. The total duration of treatment period will be 8 cycles, each lasting 3 weeks. The initial bortezomib dose is the last tolerated dose (1.0 or 1.3 milligram per metersquare [mg/ m^2] on the previous bortezomib-based treatment. Participants who start the study on a dose of 1.0 mg/m^2 bortezomib and tolerate the dose well could have their dose escalated to 1.3 mg/m^2. Doses above 1.3 mg/m^2 are not allowed. A complete cycle comprises 4 doses of bortezomib. Dexamethasone will be first introduced in Cycles 1 to 5 (i.e.dexamethasone will not be introduced for the first time in Cycles 6 to 8). The median total dose of dexamethasone received per cycle ranges from 120 mg (cycle 7) to 160 mg (cycles 1 to 6 and 8). Efficacy will be primarily assessed by determining Best Confirmed Response according to the European Group for Blood and Marrow Transplantation (EBMT) criteria. Participant's safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participant was previously diagnosed with multiple myeloma based on standard criteria and had measurable disease. Measurable disease for secretory multiple myeloma was defined as any quantifiable serum M-protein value (generally, but not exclusively, greater than (>) 1 gram per deciliter (g/dL) immunoglobulin (Ig) G Myeloma protein (M-protein) and >0.5 g/dL Ig A) or urine light-chain excretion of equal to (=) or >200 milligram (mg)/24 hour
* Participant previously tolerated 1.0 or 1.3 mg/metersquare (m^2) bortezomib alone or in combination with other agents and had complete response (CR) or partial response (PR) upon completion of bortezomib therapy
* It had been greater than or equal to (>=) 6 months since the participant's last bortezomibdose and the participant had progressive disease (PD) if prior response to bortezomib was PR or the participant had relapsed from CR
* Participant had a life expectancy >3 months
* If female, the participant was either postmenopausal or surgically sterilized or willing to use an acceptable method of birth control from screening through at least 30 days after completion of the last cycle

Exclusion Criteria:

* Participant had received chemotherapy, radiotherapy, antibody, immunotherapy, or experimental therapy to treat multiple myeloma since their last dose of bortezomib. Note: participants could have received localized palliative radiotherapy for complications due to osteolytic bone lesions. Participants could have received steroids (dexamethasone or equivalent) or thalidomide or interferon as maintenance therapy since their last dose of bortezomib according to local standard of care. In addition, participants could have received a cumulative dose of up to 160 mg dexamethasone or equivalent as emergency therapy within 4 weeks prior to enrolment. Participants could have received high dose therapy/stem cell transplantation after induction regimen containing bortezomib, but only if PR or CR was observed during bortezomib containing induction therapy
* Participant had uncontrolled or severe cardiovascular disease, including myocardial infarction within 6 months of enrolment or had New York Heart Association Class III or IV heart failure, uncontrolled angina, clinically significant pericardial disease, severe uncontrolled ventricular arrhythmias or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Participant had poorly controlled hypertension, diabetes mellitus, or other serious medical or psychiatric illness that could potentially interfere with the completion of treatment according to the protocol
* Participant had another malignancy within the past 5 years. Exceptions were made for the following if they were treated and not active: basal cell or non-metastatic squamous cell carcinoma of the skin, cervical carcinoma in situ or International Federation of Gynecology and Obstetrics Stage 1 carcinoma of the cervix
* Patient has an uncontrolled or severe cardiovascular disease, within 6 months of enrolment
* Female participant was pregnant or breast feeding. Confirmation that the participant was not pregnant was to be established by a negative beta human chorionic gonadotropin pregnancy test result obtained during the Screening period. Pregnancy testing was not required for post menopausal or surgically sterilized women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2006-06; Primary Completion 2009-02 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Best Confirmed Response to Bortezomib Re-Treatment | Day 1 of every alternate cycle starting from Cycle 1 up to End of Treatment (30 to 42 days after last dose administration of bortezomib)
  Number of participants with best confirmed response to bortezomib Re-Treatment will be assessed by the European Group for Blood and Marrow Transplantation (EBMT) criteria. Best confirmed response is, if administration of bortezomib provide continuing or additional clinical benefit after previous bortezomib administration. The ordering of possible responses are Complete Response (CR), Partial Response (PR), Minimal Response (MR), No Change (NC) and Progressive Disease (PD)/relapse from CR. CR is the best response and the poorest response is PD or relapse from CR.

SECONDARY OUTCOMES:
Participants With Percent Change in Baseline Serum Monoclonal Protein (M-protein) Best Confirmed Response Category | Day 1 of every alternate cycle starting from Cycle 1 up to End of Treatment (30 to 42 days after last dose administration of bortezomib)
  Number of participants with percent change in baseline serum M-protein best confirmed response category will be assessed by EBMT criteria. Best confirmed response is, if administration of bortezomib provide continuing or additional clinical benefit after previous bortezomib administration. Decrease in serum M-protein levels from baseline represents improvement. Participants having baseline M-protein value of <5 gram per liter (g/L) (serum) or <200 mg/24 hour (urine) will be classed in 'Not Evaluable' category and any response rate (RR) which is unconfirmed will be classed as 'Missing'.
Participants with Percent Change in Baseline Urine Monoclonal Protein (M-protein) Best Confirmed Response Category | Day 1 of every alternate cycle starting from Cycle 1 up to End of Treatment (30 to 42 days after last dose administration of bortezomib)
  Number of participants with percent change in baseline Urine M-protein best confirmed response category will be assessed by EBMT criteria. According to EBMT best confirmed response is, if administration of bortezomib provide continuing or additional clinical benefit after previous bortezomib administration. Decrease in urine M-protein levels from baseline represents improvement. Participants having baseline M-protein value of <5 g/L (serum) or <200 mg/24 hour(urine) will be classed in 'Not Evaluable' category and any RR which is unconfirmed will be classed as 'Missing'.
Duration of Best Confirmed Response (DOR) | Day 1 Cycle 1 up to last follow-up visit (8 weeks until PD)
  The DOR is defined as the duration (months) from the date of the first evidence of a best confirmed response to the date of first documented evidence of PD (or relapse for participants who experienced CR). The PD or relapse are defined as one or more of following criteria: >25% increase in either serum or urine M-protein, >25% increase in plasma cells on bone marrow, Definite increase in size of bone lesion or plasmacytoma, Development of new bone lesion or plasmacytoma, Development of hypercalcaemia. The DOR will be calculated separately in participants with a best confirmed response of >=PR.
Time to Progression (TTP) for Best Confirmed Response | (Day 1 Cycle 1 up to last follow-up visit date (8 weeks until PD)
  The TTP is defined as the duration (in months) from the date of first study treatment administration (enrollment at Day 1, Cycle 1) until the date of first documented evidence of PD (or relapse for participants who experienced CR). PD or relapse are defined as one or more of the following criteria: ->25% increase in either serum or urine M-protein. ->25% increase in plasma cells on bone marrow. -Definite increase in size of bone lesion or plasmacytoma. -Development of new bone lesion or plasmacytoma. -Development of hypercalcaemia

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (38):
- Austria (3):
  - Graz
  - Oberpullendorf
  - Vienna
- Belgium (4):
  - Antwerp
  - Brussels
  - Ghent
  - Roeselare
- France (6):
  - Dijon
  - Limousis
  - Marseille
  - Nantes
  - Paris
  - Pessac
- Germany (10):
  - Bad Soden
  - Berlin
  - Cologne
  - Erlangen
  - Hamburg
  - Hamm
  - Hanover
  - Kiel
  - Mainz
  - Würselen
- Greece (3):
  - Athens
  - Pátrai
  - Thessalonikis
- Luxembourg, Luxembourg
- Portugal (3):
  - Almada
  - Coimbra
  - Lisbon
- Spain (8):
  - Barcelona
  - Cadiz
  - Málaga
  - Salamanca
  - Santiago de Compostela
  - Seville
  - Toledo
  - Zaragoza

REFERENCES:
- See also: A Phase II, Open-label Trial Using Velcade for Re-treatment of Multiple Myeloma Subjects Following an Initial Response to Velcade. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=220&filename=CR010519_CSR.pdf